CLINICAL TRIAL: NCT00894218
Title: New Tool of Subjective and Objective Functional Evaluation and the Quality of Life After Arthroplastic Surgery of the Hip and the Knee Assisted or Not by Computer and Mini-invasive Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007-26; 2007-A0084845
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Hip Arthritis; Knee Arthritis
MeSH Terms: interventions — Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conventional arthroplasty (Active Comparator): Total hip or knee conventional arthroplasty
  Interventions: Procedure: Arthroplasty
- Mini-invasive arthroplasty (Experimental): Total hip or knee mini-invasive arthroplasty
  Interventions: Procedure: Arthroplasty
- Mini-invasive and computer-assisted arthroplasty (Experimental): Mini-invasive and computer-assisted total hip or knee arthroplasty
  Interventions: Procedure: Arthroplasty

INTERVENTIONS:
Procedure: Arthroplasty — Hip or knee arthroplasty

SUMMARY:
Hip or knee arthroplasties allow a relief of pain and a good functional habilitative at patients suffering from degenerative osteoarthritis of these articulations with medium and long-term good results. The main objective of this study is to compare the efficiency in short and medium-term functional impact parlance of two surgical techniques: computer-assisted surgery and mini-invasive surgery compared to the conventional techniques thanks to an innovative technology of ambulatory analysis of walking.

ELIGIBILITY:
Inclusion Criteria:

* Weight < 100 kg
* score UCLA > 4
* prosthesis of first intention

Exclusion Criteria:

* Pregnant
* score UCLA < 4
* osteotomy near to prosthesis
* prosthesis requiring an osseous transplant
* prosthesis already set up
* infections, contagious diseases (HIV, tuberculosis, hepatitis, venereal diseases) or metastasis
* neuromuscular diseases able to perturb walking or staying
* congenital or acquired disease, or previous surgery able to have consequences on results and prosthesis survey according to the surgeon

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To compare the efficiency in short and medium-term functional impact parlance of two surgical techniques: computer-assisted surgery and mini-invasive surgery compared to the conventional techniques | 2 years after surgery

SECONDARY OUTCOMES:
Ambulatory analysis of the walking and coordination of lower limbs, direct and indirect costs | 2 years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique-Hopitaux de Marseille, Marseille, France